CLINICAL TRIAL: NCT01987245
Title: The Application Research of Plethysmographic Waveform in Quality Control Feedback System During Cardiopulmonary Resuscitation
Brief Title: Plethysmographic Waveform for Monitoring the Quality of Cardiopulmonary Resuscitation
Acronym: PWMQC
Status: Completed | Type: Observational
Sponsor: Jun Xu (Other)
Responsible Party: Sponsor-Investigator, Jun Xu, Emergency Department, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: 2013S-512; 2011-4001-04 (Other Grant/Funding Number: CHRDS)
Record Dates: First submitted 2013-11-05; First posted 2013-11-19 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Cardiopulmonary Arrest; Cardiopulmonary Resuscitation; Return of Spontaneous Circulation; Pulse Oximeter Plethysmographic Waveform
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiopulmonary resuscitation(CPR) is the key to success for high-quality early cardiopulmonary resuscitation, and its success in the restoration of spontaneous circulation (ROSC), therefore, monitoring the quality of cardiopulmonary resuscitation and early identification ROSC is very important. Now there is no an easy, non-invasive and real-time method to monitor the quality of CPR. In this study the investigators hypothesis the pulse oximeter waveform can real-time monitor the quality of CPR ,and feedback the quality of CPR to the physicians.

ELIGIBILITY:
Inclusion Criteria:

* cardiopulmonary arrest, without do-not-resuscitation(DNR) patients
* After cardiac arrest, there is no more than 10 minutes until basic life support.
* must be carried out advanced life support (tracheal intubation and end-tidal carbon dioxide monitoring)
* comply with ethical requirements and signed informed consent

Exclusion Criteria:

* DNR patients
* rib fractures
* hemorrhagic shock caused cardiac arrest
* severe anemia, hemoglobin less than 7g/dl
* tension pneumothorax without closed drainage
* pulmonary embolism or pericardial tamponade caused cardiac arrest
* onychomycosis
* people who paint fingernails
* clearly influential peripheral oximetry underlying diseases (such as Raynaud's phenomenon, vasculitis)
* The study physicians believe there is any case is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: emergency room sample of multi-centers
Sampling Method: Non-Probability Sample
Enrollment: 617 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
survival rate | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- PUMCH, Beijing, China

REFERENCES:
- [Derived] Hu Y, Xu J, Zhu H, Zhang G, Sun F, Zhang Y, Yu X. [Profile and outcome of cardiopulmonary resuscitation after sudden cardiac arrests in the emergency department: a multicenter prospective observational study]. Zhonghua Wei Zhong Bing Ji Jiu Yi Xue. 2018 Mar;30(3):234-239. doi: 10.3760/cma.j.issn.2095-4352.2018.03.009. Chinese. PMID 29519282